CLINICAL TRIAL: NCT00657644
Title: Open-label Multi-centre Non Randomised Study of Efficacy and Safety of Vardenafil (BAY 38-9456; SB-782528) Administered in Flexible-dose Regimen in Males With Erectile Dysfunction of Broad Aetiology.
Brief Title: Efficacy and Safety of Vardenafil in Men With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11182
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 4 weeks treatment with 10 mg vardenafil followed by a flexible titration phase for 8 weeks

SUMMARY:
To find out more information on how effective and safe vardenafil is at treating impotence in men living in Russia.

ELIGIBILITY:
Inclusion Criteria:

* Males with ED according to the NIH definition (the inability to achieve or maintain penile erection sufficient for satisfactory sexual performance) for at least 3 months.
* Heterosexual relationship
* Age range: 18 years and older
* Documented written Informed Consent
* The subject must make at least four attempts at sexual intercourse (according to the question in the subject diary "Was sexual activity initiated with the intention of intercourse?") on four separate days during the untreated baseline period. At least 50% of attempts during this period must be unsuccessful, according to the following questions from the subject diary [at least one question should be answered "No"] "Were you able to achieve at least partial erection (some enlargement of the penis)?", "Were you able to insert your penis in your partner's vagina?" and "Did your erection last long enough for you to have successful intercourse?".

Exclusion Criteria:

* Any unstable medical, psychiatric, or substance abuse disorder that in the opinion of the Investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
* Presence of penile anatomical abnormalities (e.g. penile fibrosis or Peyronie's disease) that in the opinion of the Investigator would significantly impair erectile function
* Primary hypoactive sexual desire
* Spinal cord injury
* History of surgical prostatectomy (excluding TURP).
* Retinitis pigmentosa
* History of positive test for Hepatitis B surface antigen (HBsAg) or Hepatitis C.
* History of positive test for HIV.9. Severe chronic or acute liver disease, history of moderate or severe hepatic impairment.
* Clinically significant chronic hematological disease, which may lead to priapism such as sickle cell anemia and leukemia.
* Bleeding disorder.
* Significant active peptic ulceration.
* Unstable angina pectoris
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months
* Uncontrolled atrial fibrillation/flutter at screening (ventricular response rate > 100 bpm).
* Resting hypotension (a resting systolic blood pressure of < 90 mm Hg) or hypertension (a resting systolic blood pressure > 170 mm Hg or a resting diastolic blood pressure > 110 mm Hg)
* NYHA Class III and IV heart failure
* Symptomatic postural hypotension within 6 months of visit 1.
* History of malignancy within the past 5 years (other than squamous or basal cell skin cancer).

Concomitant Medication:

* Subjects who are taking nitrates or nitric oxide donors.
* Subjects who are taking anti-androgens
* Subjects who are taking androgens.
* Subjects who take anticoagulants, except for antiplatelet agents.
* Subjects who have received any investigational drug (including placebo) within 30 days of visit 1.6. Use of any treatment for ED within the 7 days of visit 1 or during the study, including oral medications, vacuum devices, constrictive devices, injections or urethral suppositories.
* Subjects who are taking the following potent inhibitors of cytochrome P- 450 3A4: HIV protease inhibitors such as ritonavir or indinavir, the anti-mycotic agents itraconazole and ketoconazole (topical forms are allowed) or erythromycin.
* Subjects who are taking alpha-blockers.

Abnormal Laboratory Values:

* Subjects who have a serum total testosterone level greater than 25% below the lower limit of normal according to the range of the testing laboratory
* Subjects with a serum creatinine >3.0 mg/dl
* Elevation of AST and/or ALT >3X the ULN.
* Diabetic subjects with an HbA1c >12%.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2003-08; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Erectile Function (EF) domain score | Week 12

SECONDARY OUTCOMES:
Erectile Function (EF) domain score | Week 4, 8 and 12 Last Observation Carried Forward (LOCF)
Change from baseline of Erectile Function domain score | Week 4, 8 and 12 Last Observation Carried Forward (LOCF)
IIEF domain scores | Week 4, 8, 12 and 12 Last Observation Carried Forward (LOCF)
Patient Diary Questions | Week 4, 8, 12 and 12 Last Observation Carried Forward (LOCF)
Global Assessment Question (GAQ) | Week 4, 8, 12 and 12 Last Observation Carried Forward (LOCF)
Premature termination, adverse events, laboratory abnormalities and concomitant medication usage | Week 4, 8 and 12
Measurements and changes from baseline in vital signs, ECG cardiac cycle measurements and ECG heart rate | Week 12
Haematology, Clinical Chemistry, Urinalysis | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Russia (2):
  - Moscow
  - Saint Petersburg